CLINICAL TRIAL: NCT02725151
Title: The Role of Inferior Vena Cava in Emergency Treatment of Acute Decompensated Heart Failure and Deciding Hospitalization
Brief Title: Acute Heart Failure Monitoring Via Inferior Vena Cava Ultrasound
Status: Completed | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Adnan Yamanoğlu, Emergency Medicine Specialist, Haseki Training and Research Hospital
Other Study IDs: 231
Record Dates: First submitted 2016-03-20; First posted 2016-03-31 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Chronic Heart Failure
Keywords: inferior vena cava ultrasound; acute; heart failure; management; decompensation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Known before diagnosed heart failure and used diuretic therapy patients will be admitted in this study.The objective of this work is whether the Inferior Vena Cava Ultrasound can be used for management of Acute Heart failure therapy. And investigators will calculation correlation of extracted urine amount with Inferior Vena Cava diameter change. Researchers will not interfere to standard recommended treatment protocol, researchers will correlated the urine amount and changed vital signs with therapy with Vena cava inferior diameter.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 years of age) of both sexes)
* Non-trauma patients
* Non- pregnant patients
* All patients will be accepted for this study, that known Heart Failure and must be taken diuretic therapy because of volume overload

Exclusion Criteria:

* Cardiac tamponade
* Aortic dissection
* Patients who had suffered cardiopulmonary arrest or been intubated

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients constitute the study population that was admitted to emergency department with complaint of dyspnea.These patients will be accepted for this study, that known Heart Failure and must be taken diuretic therapy because of volume overload.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Vena cava inferior diameter change end of each 500cc urination | Maximum 3 hours

SECONDARY OUTCOMES:
Vena cava inferior diameter change with classic treatment at each hour | Maximum 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Yamanoğlu, MD, Principal Investigator — Haseki Training and Research Hospital, Emergency Department
Locations (1):
- Adnan Yamanoğlu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Already in the nearest congress will be shared as an oral presentation or poster

REFERENCES:
- [Derived] Yamanoglu A, Celebi Yamanoglu NG, Ozturk S, Cakmak S, Akay S, Akyol PY, Sogut O. The value of the inferior vena cava ultrasound in the decision to hospitalise in patients with acute decompensated heart failure; the best sonographic measurement method? Acta Cardiol. 2021 May;76(3):245-257. doi: 10.1080/00015385.2020.1740422. Epub 2020 Mar 19. PMID 32189575